CLINICAL TRIAL: NCT03582982
Title: Flywheel Resistance Exercise to Improve Skeletal Muscle in Veterans With Chronic Kidney Disease
Brief Title: Flywheel Exercise for CKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 01903
Record Dates: First submitted 2018-06-15; First posted 2018-07-11 (Actual); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Chronic Kidney Disease stage3; Chronic Kidney Disease stage4
Keywords: resistance exercise; muscle fatigue; physical function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eccentric overload exercise (Experimental)
  Interventions: Behavioral: Eccentric overload exercise

INTERVENTIONS:
Behavioral: Eccentric overload exercise — 12 weeks of 2x per week of the following eccentric exercises: squat, shoulder press, row, and bicep curl.

SUMMARY:
Among Veterans, the prevalence of chronic kidney disease (CKD) is reported to be as high as 47.3% and a third higher than the general population. Muscle wasting and dysfunction have been identified as primary consequences of CKD. Disease-induced reductions in lean tissue adversely affect muscle fatigability. Consequently, muscle fatigability may serve as a potential limiting factor that contributes to activity limitations. However, there is a lack of evidence informing our understanding of muscle fatigability in patients with CKD. Dialysis treatment is a major factor contributing to the high financial costs of CKD care. Thus, in addition to potential health and quality of life benefits, treatments capable of maintaining kidney function or delaying the onset of dialysis treatment would provide substantial socio-economic benefit. Both lean body mass and muscle fatigability may be improved through strength training. Eccentric-overload (i.e. muscle lengthening) progressive resistance exercise (PRE) has been shown to be safe and effective for a variety of chronic conditions. Eccentric PRE using portable flywheel technology may provide a clinically viable treatment option to combat muscle impairments in CKD given the cost effectiveness and minimal space requirements for this mode of exercise.

The purpose of this study is to assess feasibility of the eccentric-overload PRE regimen for Veterans with CKD stage 3 & 4 predialysis using a prospective single-arm pre-test post-test intervention design. The primary aim of the project is to determine the effects of eccentric-overload PRE on muscle fatigability in Veterans with CKD Stages 3 & 4 predialysis. Feasibility of the regimen will be determined by the time needed to complete the 4-exercise regimen and the perceived exertion levels reported by the study participants.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory patients (with or without a gait aid)
* CKD stage 3 or 4
* patients receiving care at the DC VAMC Renal Service
* the ability to speak and read English
* orientation to person, place, and time

Exclusion Criteria:

* unable to speak English
* acute renal failure
* pregnant
* unable to follow study instructions
* any uncontrolled cardiovascular or musculoskeletal problems that would make participation in this study unsafe

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2019-02-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Knee extensor isokinetic muscle fatigability index at 12 weeks | Baseline, Week 12
  Knee extensor muscle fatigability will be assessed using a protocol consisting of 30 repetitions or to failure, whichever comes first, at their maximum strength
Change in Muscle blood flow at 12 weeks | Baseline, Week 12
  Blood flow will be assessed using Doppler ultrasound
Change in Isokinetic and isometric peak knee extension force at 12 weeks | Baseline, Week 6, Week 12
  Unilateral peak knee extension/flexion isokinetic force (at 180º/s and 60º/s) will be obtained across five continuous repetitions using a load cell
Change in Short Physical Performance Battery at 12 weeks | Baseline, Week 12
  This composite score is made up of measures of balance, gait speed (15 ft), and timed chair stands (x5).
Change in Timed Up-and-Go at 12 weeks | Baseline, Week 12
  This test will begin the test with the subject fully sitting in a chair with arm rests, with the upright mobility portion of the test focused on an easily visible marked target 3 meters away from the chair
Change in Lean Body Mass, as estimated by diagnostic ultrasound at 12 weeks | Baseline, Week 6, Week 12
  Sonographic estimates of LBM (aggregate muscle thickness, cm) will serve as a proxy measure for muscle tissue composition in this study
Change in myosteatosis, as estimated by diagnostic ultrasound at 12 weeks | Baseline, Week 6, Week 12
  Sonographic estimates of myosteatosis (grayscale, or GSL, values, 0-255) will serve as a proxy measure for muscle tissue composition in this study

SECONDARY OUTCOMES:
Change in Grip strength at 12 weeks | Baseline, Week 12
  This measure will be obtained with a hand grip dynamometer using the mean value of 3 trials under standardized conditions.
Change in Activities-Specific Balance Confidence (ABC) Scale at 12 weeks | Baseline, Week 12
  mobility questionnaire; range 0-100, with higher values indicating higher confidence
Change in Short Form Health Survey (SF-36) Scale at 12 weeks | Baseline, Week 12
  general physical functioning questionnaire; each of eight sections range 0-100 with higher values indicating less disability. The eight sections include vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health.
Change in Falls Efficacy Scale (FES) at 12 weeks | Baseline, Week 12
  fall avoidance behavior questionnaire; range 10-100, with lower values indicating greater efficacy
Change in weight at 12 weeks | Baseline, Week 6, Week 12
  Weight (in lbs) using bioelectric scale
Change in height at 12 weeks | Baseline, Week 6, Week 12
  Height (in inches) using stadiometer
Change in body water at 12 weeks | Baseline, Week 6, Week 12
  Body water (%) using bioelectric scale
Change in Blood Pressure at 12 weeks | Baseline, Week 12
  After sitting quietly for 5 minutes, resting blood pressure will be recorded in triplicate

CONTACTS AND LOCATIONS:
Overall Officials: Michael O Harris-Love, DSc, Principal Investigator — Washington DC VA Medical Center
Locations (1):
- Washington DC VA Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No